CLINICAL TRIAL: NCT05744856
Title: Living Together With Chronic Disease: Informal Support for Diabetes Management in Vietnam (VALID) - Gestational Diabetes in Vietnam - Phase II
Brief Title: A Co-created Self-care and Informal Support Intervention Study Among Women With GDM in Vietnam
Acronym: VALID-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thai Binh University of Medicine and Pharmacy (Other)
Collaborators: University of Copenhagen (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Thanh Duc Nguyen, Head of International Relations Department, Thai Binh University of Medicine and Pharmacy
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VALID II
Record Dates: First submitted 2022-12-21; First posted 2023-02-27 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: GDM
Keywords: GDM; Co-creation; Self-care; Vietnam; Low-and-middle-income countries; Informal support; Intervention
MeSH Terms: interventions — Self Care

STUDY DESIGN:
Intervention Model Description: The study is parallel 2-arm non-randomized intervention study with a delayed-start for the intervention group. The study population will be recruited in two phases. Over a period of 4 months (phase I) 1000 pregnant women will be screened for GDM among which 200 will be diagnosed with GDM and receive standard GDM care according to national guidelines in Vietnam (control group). During phase I, the "self-care + informal support intervention" will be co-created with local health care staff and a sub-group of the control group. Four months after the recruitment for phase I has finished, recruitment for phase II will start. Over a period of 4 months, another 1000 pregnant will be screened for GDM among which 200 will be diagnosed with GDM. These 200 women will be invited to receive the "self-care + informal support" intervention (intervention group). This pilot study is designed to inform a power calculation and logistics of a future full-scale randomized controlled trial.
Masking Description: Due to the overt nature of the intervention, it is not possible to blind the participants, healthcare providers nor the investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard GDM care (No Intervention): After being diagnosed with GDM, standard care includes counseling on nutrition and physical activity. All patients are referred to an endocrinologist at the General Hospital, yet this is not covered by insurance unless the patients have received a referral letter from a health station. The endocrinologist will perform blood glucose measurements (venous blood sample) once every four weeks at the General Hospital until gestational week 36, after which it will be monitored once a week until delivery. The cut-off for c-section is 3800g (no matter the mother's GDM status).
  Treatment recommended by the endocrinologist may include home-monitoring of blood glucose and insulin treatment in the most severe cases. The home-monitoring requires that the women are able to buy the glucometer and test strips themselves.
- Self-care with informal support (Experimental): Standard care + "Self-care/informal support" intervention
  The detailed content of the "self-care/informal support intervention" will be developed at participatory co-creation workshops involving pregnant women with GDM, their informal support persons, and health care staff.
  It is expected that intervention will include educational pamphlets regarding GDM and digital GDM education through videos and text messages. Further, digital coaching will be conducted and networking among intervention participants via the Vietnamese messaging app Zalo. In addition, each woman will be invited to include one informal support person in the intervention activities.
  GDM education will concern coaching on diet and exercise during pregnancy and after delivery and coaching on breastfeeding and infant/child nutrition.
  Interventions: Behavioral: Self-care with informal support

INTERVENTIONS:
Behavioral: Self-care with informal support — The detailed content of the "self-care with informal support intervention" will be developed at participatory co-creation workshops involving pregnant women with GDM, their informal support persons, and health care staff.
  It is expected that intervention will include educational pamphlets regarding GDM and digital GDM education through videos and text messages. Further, digital coaching will be conducted and networking among intervention participants via the Vietnamese messaging app Zalo. In addition, each woman will be invited to include one informal support person in the intervention activities.
  GDM education will concern coaching on diet and exercise during pregnancy and after delivery and coaching on breastfeeding and infant/child nutrition.
  Arms: Self-care with informal support

SUMMARY:
Gestational Diabetes Mellitus (GDM) is significant public health problem in Vietnam, which is potentially treatable if managed properly by the pregnant women once diagnosed. However, systematic screening for GDM is rarely undertaken in Vietnam, and little is known about how health providers, pregnant women, and their families in today's Vietnam handle the condition. Vietnamese women often depend on their extended family for daily life management and access to social and financial resources, hence, an intervention that focuses on informal support and GDM self-care may increase adherence the standard guidelines among pregnant women with GDM in Vietnam and increase neonatal and maternal health outcomes.

DETAILED DESCRIPTION:
Background: Across the globe, diabetes mellitus is attaining epidemic proportions, with low- and middle-income countries confronting particularly high burdens. VALID II focuses on gestational diabetes mellitus (GDM), a transitory form of diabetes that presents during pregnancy.

Objectives: To: i) Determine prevalence and risk factors for GDM among pregnant women in Vietnam's Thai Binh province, ii) Measure the associations between GDM and pregnancy complications and outcomes, iii) Understand how pregnant women with GDM and their informal support persons perceive and handle the condition, iv) Co-create, implement, and assess the feasibility of a intervention aiming to enhance the self-care capacities of pregnant women with GDM.

Study setting: Thai Binh, Vietnam

Study design: Intervention study

Study population: 2,000 pregnant women attending antenatal care.

Methodology: The study will be performed as a pilot parallel 2-arm non-randomized intervention study with a delayed-start for the intervention group. 1000 women will be invited into the study at their first antenatal care visit (gestational week 12) and complete a questionnaire (inclusion questionnaire). All women will be offered a 2-hour oral glucose tolerance test (OGTT) in gestational week 24-28 and complete second questionnaire (OGTT questionnaire) exploring living conditions, lifestyle, risk factors, selfcare, perceived social support, perceived wellbeing, and sign of depression. An estimated 200 women (~20%) will screen positive for GDM by the OGTT according to the World Health Organization (WHO) 2013 diagnostic criteria and receive standard GDM care. These 200 women will serve as the study's control group (study phase I). Among the 200 women who screen positive in phase I, ethnographic interviews will be formed in a subgroup of 20 women. The information from the 20 ethnographic interviews and the 200 questionnaire interviews will help inform a co-created "self-care and informal support" intervention. Subsequently, another 1000 women will be invited into the study at their first antenatal care visit and be offered a 2-hour oral glucose tolerance test (OGTT) in gestational week 24-28 (study phase II). An estimated 200 women (~20%) will screen positive for GDM, and these women will receive the co-created intervention and serve as the study's intervention group.

Additionally, all women (both intervention and control group) will be interviewed in gestational week 32-36 and 8-12 weeks postpartum. Further, information about HbA1c, maternal BMI, gestational weight gain, mode of delivery, neonatal weight as well as obstetric and neonatal complications will be obtained from measurements and the delivery records. The primary endpoint will be large for gestational age. Secondary neonatal endpoints will be macrosomia, preterm birth, stillborn/neonatal death and neonatal hypoglycemia. Secondary maternal outcomes will be HbA1c, hypertensive disorders, gestational weight gain, caesarean section, women's GDM self-care, perceived social support, perceived wellbeing, signs of depression, breastfeeding rates, quality of life, and empowerment. The outcome of this intervention pilot study will determine whether the intervention can be feasibly delivered within the context of a full-scale randomized controlled trial (RCT). Thus, the pilot study will not be powered to detect statistical differences in key clinical outcomes, but the sample sizes have been chosen to highlight problems and confirm the potential to detect differences.

Women may be included in the study all the way up to gestational age 28 depending on when they attend their first antenatal care appointment and receive the OGTT. Further, the point in time of the different questionnaire interviews may vary according to the needs of the pregnant women and when she delivers.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy < 28 weeks
* Singleton and multiple pregnancies
* Residing in Thai Binh province
* Speaks and reads Vietnamese
* Agree to participate voluntarily (informed consent)

Exclusion Criteria:

* Pre-gestational diabetes (type I or type II)
* Severe chronic disease

Women with GDM in a prior pregnancy are eligible for inclusion into the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 435 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thanh Duc Nugyen, MD, Principal Investigator — Thain Binh Medical University
Locations (2):
- Vietnam (2):
  - Thai Binh Maternity Hospital, Thái Bình, Thai Binh
  - Kim Ngan Clinic, Thái Bình, Thái Bình

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the articles will be shared after de-identification (text, tables, figures, and appendices). Sharing of data must adhere to the General Data Protection Regulation (GDPR) in Denmark and Vietnam.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be available immediately following publication. No end date.
Access Criteria: All requests for data should be addressed to the sponsor (see contact details under central contact person). The sponsor will will review the request and involve all applicable parties in the decision-making outcome (i.e. all Vietnamese and Danish collaborators). Data will be shared with researchers who provide a methodological sound proposal. New projects that result in data sharing should meet the high standards (quality, ethical, and financial) maintained by this study.

REFERENCES:
- [Derived] Linde DS, Le HM, Vu DTK, Dang NT, Nguyen AT, Vu TP, Nguyen XB, Nguyen CD, Meyrowitsch DW, Sondergaard J, Vinter CA, Bygbjerg IC, Rasch V, Nguyen TD, Gammeltoft TM, Nguyen DK. A co-created self-care and informal support intervention targeting women with gestational diabetes mellitus in northern Vietnam (VALID-II): a protocol for a two-arm non-randomised feasibility study. Pilot Feasibility Stud. 2025 May 29;11(1):73. doi: 10.1186/s40814-025-01657-x. PMID 40442746

RESULTS

PARTICIPANT FLOW:
Groups:
- Self-care With Informal Support: Standard care + "Self-care/informal support" intervention
  The women in the intervention group will receive standard care and the self-care/informal support intervention.
  The "self-care/informal support intervention" will be developed at participatory co-creation workshops involving women with GDM, their informal support persons, and health care staff.
  The intervention will include educational pamphlets regarding GDM and digital GDM education through videos and text messages. Further, digital coaching will be conducted and networking among intervention participants via the Vietnamese messaging app Zalo. In addition, each woman will be invited to include one informal support person in the intervention activities.
  GDM education will concern coaching on diet and exercise during pregnancy and after delivery and coaching on breastfeeding and infant/child nutrition.
Period: Overall Study
Arm/Group | Standard GDM Care | Self-care With Informal Support
Started (All participants assigned to each group at the STARTED milestone were women who met the eligibility criteria outlined in the study protocol.) | 233 | 202
Completed (Women who were lost to follow up were excluded at the COMPLETED milestone) | 230 | 199
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Population: Numbers of participants assigned to the arms in Participant Flow are number of women who satisfied the eligible criteria indicated in the Protocol in clinicaltrials.gov. Those numbers are larger than the numbers reported in Baseline Measures because women with twin gestation were excluded. This exclusion was necessary to preserve the validity of our primary outcome analysis-large for gestational age
Groups:
- Self-care With Informal Support: Standard care + "Self-care/informal support" intervention
  The detailed content of the "self-care/informal support intervention" will be developed at participatory co-creation workshops involving pregnant women with GDM, their informal support persons, and health care staff.
  It is expected that intervention will include educational pamphlets regarding GDM and digital GDM education through videos and text messages. Further, digital coaching will be conducted and networking among intervention participants via the Vietnamese messaging app Zalo. In addition, each woman will be invited to include one informal support person in the intervention activities.
  GDM education will concern coaching on diet and exercise during pregnancy and after delivery and coaching on breastfeeding and infant/child nutrition.
  Self-care with informal support: The detailed content of the "self-care with informal support intervention" will be developed at participatory co-creation workshops involving pregnant women with GDM, their informal support persons, and health care staff.
- Total: Total of all reporting groups
Arm/Group | Standard GDM Care | Self-care With Informal Support | Total
Number analyzed (Participants) | 226 | 201 | 427
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 226 | 201 | 427
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (5.5) | 30.2 (5.2) | 30.6 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 226 | 201 | 427
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 226 | 201 | 427
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Vietnam | 226 | 201 | 427
Prepregnancy BMI [Mean (Standard Deviation); unit: kg/m2] — Pre-pregnancy body mass index (kg/m2) of enrolled women.
  kg/m2 | 21.2 (2.5) | 21.4 (2.8) | 21.3 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Large for Gestational Age (LGA)
Description: Number of Participants who delivered newborns with birth weight above or equal to the 90th percentile according to gender and gestational age based on the INTERGROWTH-21st birthweight chart
Time Frame: Delivery (up to study month 7 after enrolment/Gestational age 40)
Population: Numbers of Participants reported here are smaller than those reported in the Participant Flow because for the outcome of large-for-gestational age, participants who lost to follow up or had stillbirth were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard GDM Care | Self-care With Informal Support
Number analyzed (Participants) | 222 | 198
Participants | 23 | 17

2. Primary Outcome: Large for Gestational Age (LGA)
Description: Number of Participants who delivered newborns with birth weight above or equal to the 90th percentile according to gender and gestational age based on the INTERGROWTH-21st fetal weight formula.
Time Frame: Delivery (study month 7 after enrolment/Gestational age 40)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard GDM Care | Self-care With Informal Support
Number analyzed (Participants) | 222 | 198
Participants | 30 | 19

3. Primary Outcome: The Feasibility of the Self-care Intervention [Recruitment]
Description: Number of Participants eligible for the study who accepted to be included in the intervention arm.
Time Frame: Recruitment (study month 0)
Population: Number of Participants reported here were women who eligible for the intervention in the self-care with informal support.
Measure: Count of Participants; unit: Participants
Arm/Group | Self-care With Informal Support
Number analyzed (Participants) | 202
Participants | 202

4. Primary Outcome: The Feasibility of the Self-care Intervention [Retention]
Description: Number of Participants included in the self-care intervention group who completed the study (delivery data and post-partum interview).
Time Frame: Recruitment to post-partum evaluation (study month 0-10)
Measure: Count of Participants; unit: Participants
Arm/Group | Self-care With Informal Support
Number analyzed (Participants) | 202
Participants | 156

5. Primary Outcome: The Acceptability of the Self-care Intervention
Description: Acceptability will be measured in a combined quantitative and qualitative study. It will be measured quantitatively via 5-point likert scales among the intervention group [Range: 1-5; Minimum score: 1; Maximum score: 5; Higher score indicates high acceptability]. It will be assessed qualitatively among a sub-group of the intervention group through a ethnographic study.
Time Frame: Study month 3 to 10 /Gestational age 24 to 12 weeks post-partum
Population: The numbers of participants here were participant who provided responses of acceptability at post-partum interview.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Self-care With Informal Support
Number analyzed (Participants) | 106
score | 3.9 (0.7)

6. Secondary Outcome: Mode of Delivery
Description: Number of participants with spontaneous vaginal delivery, assisted vaginal delivery, planned c-section or emergency c-section
Time Frame: Delivery (study month 7/Gestational age 40)
Population: Number of participants reported here were women with singleton pregnancy and therefore are smaller than the numbers assigned in the Participant Flow.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard GDM Care | Self-care With Informal Support
Number analyzed (Participants) | 226 | 201
Participants
  Number of Participants who had vaginal delivery | 77 | 68
  Number of Participants who had C-section delivery | 138 | 124
  Number of Participants with missing data | 11 | 9

7. Secondary Outcome: Pre-term Birth Below Gestational Age 37+0
Description: Number of participants with spontaneous preterm birth or medical induced preterm birth
Time Frame: Delivery (study month 7/Gestational age 40)
Reporting Status: Not Posted

8. Secondary Outcome: Gestational Age
Description: The gestational age of newborns at delivery
Time Frame: Delivery (study month 7/Gestational age 40)
Reporting Status: Not Posted

9. Secondary Outcome: Birth Weight
Description: Birth weight of newborns measured in grams
Time Frame: Delivery (study month 7/Gestational age 40)
Reporting Status: Not Posted

10. Secondary Outcome: Macrosomia
Description: Number of newborns with birth weight above 4000g
Time Frame: Delivery (study month 7/Gestational age 40)
Reporting Status: Not Posted

11. Secondary Outcome: Macrosomia (Vietnam)
Description: Number of newborns with birth weight above 3500g
Time Frame: Delivery (study month 7/Gestational age 40)
Reporting Status: Not Posted

12. Secondary Outcome: Live-born
Description: Newborns that are live-born (Yes/no)
Time Frame: Delivery (study month 7/Gestational age 40)
Reporting Status: Not Posted

13. Secondary Outcome: Small for Gestational Age (SGA)
Description: Number of newborns below the 10th percentile for birth weight according to gestational age
Time Frame: Delivery (study month 7/Gestational age 40)
Reporting Status: Not Posted

14. Secondary Outcome: Apgar Score
Description: The Apgar score of newborns measured 1 and 5 minutes after delivery (score: 0-10)
Time Frame: Delivery (study month 7/Gestational age 40)
Reporting Status: Not Posted

15. Secondary Outcome: Neonatal Hypoglycemia
Description: Measurement of blood glucose (mmol/l) in newborns
Time Frame: Delivery (study month 7/Gestational age 40)
Reporting Status: Not Posted

16. Secondary Outcome: Maternal Gestational Weight Gain
Description: Change in delta weight (kilogram) among participants between gestational age 36 minus first measured/pre-gestational weight
Time Frame: Study month 0 and 6/Gestational age 12 and 36
Reporting Status: Not Posted

17. Secondary Outcome: HbA1c
Description: Change in delta score among participants between gestational age 24 and 40 (delivery)
Time Frame: Study month 3 and 7/Gestational age 24 and 40 (delivery)
Reporting Status: Not Posted

18. Secondary Outcome: Breast Feeding Practices
Description: Participants' breast feeding practices measured through ad hoc developed questions
Time Frame: Study month 10 (12 weeks post-partum)
Reporting Status: Not Posted

19. Secondary Outcome: Post-partum Depression
Description: Change in delta score among participants measured through the Edinburgh postpartum depression scale (EPDS) [10 items on 4-point scale ranging from 0-3]
Time Frame: Study month 3 and 10/Gestational age 24 and 12 weeks postpartum
Reporting Status: Not Posted

20. Secondary Outcome: Perceived Social Support
Description: Change in delta score among participants measured through the Multidimensional Scale of Perceived Social Support scale (MSPSS) [11 item 7-point scale ranging from 1-7]
Time Frame: Study month 3,6 and 10/Gestational age 24, 36 and 12 weeks postpartum
Reporting Status: Not Posted

21. Secondary Outcome: Well-being
Description: Change in delta scores measured through WHO 5 Wellbeing index [5 items on 6-point scale ranging from 0-5]
Time Frame: Study month 0, 3, 6 and 10/Gestational age 12, 24, 36 and 12 weeks postpartum
Reporting Status: Not Posted

22. Secondary Outcome: Self-care Agency
Description: Difference in score between intervention and comparator group measured through the Self-care Agency Scale-Revised (ASAS-R) [15 items on 5-point scale ranging from 1-5]
Time Frame: Study month 3 and 6/Gestational age 24 and 36
Reporting Status: Not Posted

23. Secondary Outcome: Self-care of GDM
Description: Difference in score between intervention and comparator group measured through the Summary of Diabetes Self- Care Activities (SDSCA) [10 items on 8-point scale ranging 0-7]
Time Frame: Study month 6/Gestational age 36
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Diet
Description: Change in diet measured through ad hoc developed questions
Time Frame: Study month 3 and 6/Gestational age 24 and 36
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Physical Activity
Description: Change in physical activity measured through ad hoc developed questions
Time Frame: Study month 3 and 6/Gestational age 24 and 36
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Episiotomy
Description: Number of participants where episiotomy is performed during delivery
Time Frame: Delivery (study month 7/Gestational age 40)
Reporting Status: Not Posted

27. Other Pre Specified Outcome: PPROM
Description: Number of participants with Premature Primary Rupture of Membranes
Time Frame: Delivery (study month 7/Gestational age 40)
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Prevalence of GDM
Description: Number of participants with GDM diagnosed according to WHO criteria
Time Frame: Study month 3/Gestational age 24
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Risk Factors of GDM
Description: Number of pre-gestational and gestational risk factors for GDM prevalent among participants diagnosed with GDM (risk factor are defined as according to those known in the literature, e.g. age, BMI, family disposition, gestational weigh gain)
Time Frame: Study month 3/Gestational age 24
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Perception of GDM
Description: Ethnographic study conducted among approximately 40 pregnant women with GDM and their informal support persons (20 from intervention group and 20 from control group)
Time Frame: Study month 3 to 7/Gestational age 24 to 40 (delivery)
Reporting Status: Not Posted

31. Other Pre Specified Outcome: GDM Self-care Practices
Description: as for outcome 30
Time Frame: Study month 3 to 7/Gestational age 24 to 40 (delivery)
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Perception of "Self-care/Informal Support" Intervention
Description: Ethnographic study conducted among approximately 20 pregnant women with GDM and their informal support persons (intervention group)
Time Frame: Study month 3 to 10/Gestational age 24 to 12 weeks post-partum
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Family Health
Description: The short form version of the Family Health Scale [10 items on a 5-point scale ranging from 1-5]. A total score of 0-5 indicates poor family health, 6-8 indicates moderate family health, and 9-10 indicates excellent family health
Time Frame: Study month 6/Gestational age 36
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Costs
Description: Direct economic costs (in Vietnamese Dong/VND and USD) and indirect costs (human ressources measured in hours) spent on developing the intervention
Time Frame: Throughout whole study (study month 0-10)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the period from diagnosis of GDM to delivery, an average of 3 months
Arm/Group | Standard GDM Care | Self-care With Informal Support
All-Cause Mortality (participants affected / at risk) | 0/223 | 0/198
Serious Adverse Events (participants affected / at risk) | 0/223 | 0/198
Other Adverse Events (participants affected / at risk) | 0/223 | 0/198

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT05744856/Prot_SAP_000.pdf